CLINICAL TRIAL: NCT06676423
Title: A Phase I Clinical Trial to Evaluate the Safety of Neuronata-R® Inj. Suspended With HypoTHermosol® FRS (HTS-FRS) in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Evaluate the Safety of Neuronata-R® Inj. Suspended With HypoTHermosol® FRS (HTS-FRS) in Patients With ALS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corestemchemon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEURONATA-ALSHT122
Record Dates: First submitted 2024-06-16; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Mesenchymal stem cell; cell theraphy; ALS; HypoThermosol(HTS-FRS); Phase 1 clinical trial
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Riluzole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Groups/Cohorts (Experimental): In the first-stage dose, a 1:1 mixture of autologous CSF and HypoThermosol® FRS (HTS-FRS) is used as a suspension, and in the second-stage dose, only HypoThermosol® FRS (HTS-FRS) is used as a suspension without cerebrospinal fluid.
  Mix 1.0 ⅹ 10^6 cells per kg of body weight with the suspension at the dose level below
  1. First stage dose: HTS-FRS 0.5mL/10kg + cerebrospinal fluid 0.5mL/10kg
  2. Second stage dose: HTS-FRS 1.0mL/10kg
  Interventions: Biological: Lenzumestrocel; Drug: Riluzole

INTERVENTIONS:
Biological: Lenzumestrocel — 1.0 ⅹ 10^6 cells/kg of Neuronata-R mixed with HTS-FRS suspension are administered twice in the cerebrospinal fluid at intervals of 26 days
  Other Names: Neuronata-R; Autologous Bone Marrow derived Mesenchymal Stem cell
Drug: Riluzole — In the case of a subject who is not taking Riluzole at the time of screening (visit 1), Riluzole should be taken except when discontinued due to Adverse events. The dose can be changed within the authorization according to the medical expert's judgement
  Other Names: Rilutek

SUMMARY:
This clinical trial is a single-center, open-label, and phase I clinical trial to Evaluate the Safety of Neuronata-R® Inj. suspended with HypoTHermosol® FRS (HTS-FRS) in Patients with Amyotrophic Lateral Sclerosis.

DETAILED DESCRIPTION:
Neuronata-R is produced by mixing the patient's own cerebrospinal fluid with cultured mesenchymal stem cells the day before administration. Therefore, as autologous cerebrospinal fluid is collected from the patient for drug production at each administration, the patient must endure the occurrence of adverse events (headache, pain, etc.) and pain caused by collection, and problems such as fatigue and time consumption of the medical staff's procedure have continuously emerged.

Therefore, a comparative equivalence tests and stability tests were conducted with HypoThermosol® FRS (HTS-FRS) as a suspension agent for Neuronata-R, and it was confirmed that there was no difference in the quality of the finished product depending on the type of additive and Neuronata-R using autologous cerebrospinal fluid as a suspension agent, and it was confirmed that it was safe as an additive through non-clinical trials.

The dose determination for the safety evaluation of HypoThermosol® FRS (HTS-FRS), which will be used as a suspension, was determined in consultation with the MFDS to use a 1:1 mixture of autologous CSF and HypoThermosol® FRS (HTS-FRS) as a suspension in the first stage dose, and only HypoThermosol® FRS (HTS-FRS) was used as a suspension in the second stage dose without cerebrospinal fluid. And, the administration period is follow-up for 4 weeks after administration twice every 26 days.

ELIGIBILITY:
Inclusion Criteria:

1. Among subjects diagnosed with familial or sporadic amyotrophic lateral sclerosis
2. Subjects whose ALSFRS-R scores are in the range of 25~46 at the time of screening (Visit 1).
3. Subjects who are able to visit the site by themselves or with other's support.
4. When subjects and/or their legal guardians consent to participating in this clinical study.
5. Subjects deemed, by the investigator, capable of complying with the clinical study protocol
6. For child-bearing aged female subjects: Subjects who consent to sexual abstinence (refraining from sexual intercourse) or use of contraception method with annual failure rate of < 1% during the study period.

A female subject who has experienced the menarche, does not reach the menopause (or 12-month or longer amenorrhea for unknown reasons except menopause) and does not receive surgical sterilization (ovariectomy and/or hysterectomy) is regarded as the child-bearing aged woman.

Examples of contraception methods with annual failure rate of < 1% include bilateral tubal ligation, vasectomy, appropriate use of hormonal contraceptives that inhibit ovulation (supplemented by barrier method and spermicide), hormone-releasing intrauterine device and copper intrauterine device.

Based on clinical study period and subject's preferred lifestyle, the reliability of sexual abstinence should be evaluated. Periodic abstinence (e.g., calendar method, ovulation and post-ovulation symptothermal method) and extravaginal ejaculation are not acceptable contraception methods.

For male subjects: Subjects who, as described below, consent to sexual abstinence (refraining from sexual intercourse) or use of contraception method and consent to refrain from donation of sperm.

When a male subject has his child-bearing aged female partner or pregnant female partner, he should maintain sexual abstinence or use condom to avoid exposure to embryo. Such male subject should not donate sperm during this period.

Based on clinical study period and subject's preferred lifestyle, the reliability of sexual abstinence should be evaluated. Periodic abstinence and extravaginal ejaculation are not acceptable contraception methods.

Exclusion Criteria:

1. Subjects who fail to satisfy ALS diagnosis criteria according to the revised World Federation of Neurology El Escorial Criteria [Rix Brooks, 2000].
2. Subjects expected to have side effects on administration of cell therapy (such as subjects suspected to have malignant tumor, high-risk subjects vulnerable to psychogenic shock and severe hypertension subjects).
3. ALSFRS-R score of less than 25 and 47 or higher during screening (visit 1)
4. Subjects who fall into above Class II according to the New York Heart Association's functional classification (see the attachment), who have showed myocardial infarction, unstable arrhythmia and/or other significant cardiovascular diseases such as unstable angina in the past 3 months, or who show electrocardiographic signs of myocardial infarction or angina at the time of screening (Visit 1) or who received stent insertion or coronary artery bypass grafting.
5. Subjects who have experienced epileptic seizure.
6. Subjects with severe renal disorder (serum creatinine: not less than 3.0 mg/dL).
7. Subjects with severe hepatic disorder (ALT, AST, or bilirubin: over 2.0 times of the normal upper limit).
8. Subjects who show hemorrhagic tendency at the time of screening (PT and aPTT > 1.5 x ULN)
9. Subjects who are found to have active viral infections (such as HBsAg, HCV Ab, HIV Ab, CMV IgM, EBV IgM, HSV IgM and Treponema pallidum) at the time of screening.
10. Subjects with hypersensitivity to antibiotics (penicillin or streptomycin).
11. Subjects with any malignant tumor in the past 5 years before screening, except malignant tumors with very low risk of metastasis or death (such as appropriately treated cervical intraepithelial neoplasia, skin basal or squamous cell carcinoma, localized prostate cancer or ductal carcinoma in situ).
12. Subjects who are receiving any medicinal products that may affect bone marrow functions.
13. Subjects with severe mental disorders (such as schizophrenia and bipolar disorder. However, exception applies to mild ALS-related cognitive impairment and secondary emotional trauma).
14. Subjects for whom administration of investigational product is prohibited, subjects with conditions that may affect interpretation of results or subjects with conditions that may result in high risk of complications, such as the rest diseases, metabolic disorders, physical examination results and/or laboratory test results as diseases or such conditions are reasonably suspected.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
tolerability Assessment | through study period, an average of 8week
  HTS-FRS DLT expression for each dose step
Safety Assessment | through study period, an average of 8week
  Adverse Events(including DLT)
Safety Assessment | Baseline and 26day, 8week
  Clinical Laboratory Analysis(Change in laboratory test results at the time of visit after IP administration compared to baseline)
Safety Assessment | 0 Day, 26 Day
  Cerebrospinal Fluid Analysis(Changes in cerebrospinal fluid results at 26day compared to 0day)

SECONDARY OUTCOMES:
Exploratory Assessment | baseline and 26day , 8week
  Change in total ALSFRS-R score from before treatment (screening) to after administration
Exploratory Assessment | within -8week and 0day, 8week
  Change rate in ALSFRS-R score from before treatment (screening) to after administration

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyun Kim, MD, PhD, Principal Investigator — Hanyang University Seoul Hospital
Locations (1):
- Hanyang university hospital, Seoul, South Korea